CLINICAL TRIAL: NCT06004713
Title: Multi-center, Non-interventional, Prospective Registry Study on the Treatment of Solid Tumors With Mismatch Repair Deficiency or Microsatellite Instability
Brief Title: Registry Study in MSI/dMMR Solid Tumors
Status: Recruiting | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Other Study IDs: LGH2023093
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-07

CONDITIONS: DMMR Cancer; MSI-H; Solid Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Blood sample collection: Collect 10mL of peripheral blood in a purple EDTA-K2 anticoagulant blood collection tube. If the blood plasma cannot be separated within the specified time, a Streck (EDTA-K3) blood collection tube can be used, and the patient's name, sample type, and collection time should be marked on the tube wall.
  2. Plasma Separation: Whole blood samples are centrifuged at 4°C or room temperature, at 1800g for 10 minutes. Except for 0.5mL of whole blood reserved, all the whole blood is separated into plasma as much as possible. After centrifugation, carefully collect the upper layer of plasma into a new, labeled 5mL low-adsorption centrifuge tube, and finally seal with a sealing film for future use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort A: Patients will initially receive monotherapy PD1/PDL1 monoclonal antibody therapy.
- Cohort B: Patients will initially receive dual blockade of both PD1/PDL1 and CTLA4
- Cohort C: Patients will initially receive PD1/PDL1 monoclonal antibody combined with chemotherapy or targeted therapy.
- Cohort D: Patients will receive other standard treatments for this tumor other than ICIs.

SUMMARY:
This study is a multi-center, non-interventional, prospective clinical observational study, aiming to evaluate the effectiveness and safety of subsequent treatment in dMMR/MSI solid tumor patients who have never received ICIs under real-world conditions. Particular attention is paid to the efficacy in populations where treatment plans are adjusted based on ctDNA, and potential predictive or prognostic biomarkers are explored.

DETAILED DESCRIPTION:
This study plans to enroll patients in the following four cohorts:

* Cohort A: Initially only receiving PD1/PDL1 monotherapy;
* Cohort B: Initially receiving simultaneous blockade of PD1/PDL1 and CTLA4;
* Cohort C: Initially receiving PD1/PDL1 monotherapy combined with chemotherapy or targeted therapy;
* Cohort D: Initially not using ICIs, receiving other standard treatments for this tumor type

To explore the role of ctDNA testing in therapeutic decision-making, patients with the first evaluation of SD in cohort A are divided into two groups: ctDNA testing/intervention group (Group A1) and ctDNA testing/non-intervention group (Group A2). In group A1, if there is no early response to ctDNA, the researchers and the patient will decide to add CTLA4 antibody or other potentially effective treatments after thorough communication. If there is an early response to ctDNA, then continue with PD1/PDL1 monoclonal antibody treatment. Patients in group A2 undergo ctDNA testing, but still continue with PD1/PDL1 monoclonal antibody treatment according to the RECIST v1.1 standard when the first evaluation of SD is made. Meanwhile, explore the role of 1-year ctDNA-MRD in guiding treatment in patients with long-term tumor control, and explore the guiding role of re-biopsy of tumor tissue or ctDNA testing in helping making treatment regimen after progression on ICIs.

Number of Subjects:

• This study will recruit patients nationwide for data collection over a period of 3 years. The plan is to enroll 100 cases in Cohort A, including 25 cases in Group A1 and 25 cases in Group A2; 30 cases in Cohort B; 30 cases in Cohort C; and 30 cases in Cohort D.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form and voluntarily participate in this study;
* Age ≥ 18 years old; age should also be ≤75 years old in Cohorts B, C, D;
* Histologically or cytologically confirmed to have a solid malignant tumor and confirmed by immunohistochemistry to be dMMR or confirmed by PCR/NGS to be MSI;
* The researcher determines that the patient can receive anti-tumor treatment;
* Have evaluable lesions

Exclusion Criteria:

* Other malignant tumors within 5 years before joining the study, except for cured skin squamous cell carcinoma, basal cell carcinoma, non-muscle invasive bladder cancer, localized low-risk prostate cancer (defined as stage ≤T2a, Gleason score ≤6 points, and prostate cancer diagnosed with PSA ≤10 ng/mL (if measured). Patients who have received radical treatment and have no prostate specific antigen (PSA) biochemical recurrence can participate in this study), cervical/breast carcinoma in situ, and Lynch syndrome;
* Evidence already exists that the patient is a pregnant or lactating woman;
* Previous treatment with immune checkpoint inhibitors or T cell co-stimulatory drugs, including but not limited to PD1, CTLA4, LAG3, and other immune checkpoint blockers, therapeutic vaccines, etc.; patients exposed to ICIs in perioperative setting are allowed to be enrolled if disease relapse after more than 6 months since the last dose of ICIs;
* Other situations deemed by the researcher to be unsuitable for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The estimated start time of this study is August 2023, and data will be collected from enrolled patients nationwide over a period of 3 years. It is planned to enroll 100 patients in Cohort A, including 25 in Group A1 and 25 in Group A2. It is planned to enroll 30 patients in Cohort B, 30 in Cohort C, and 30 in Cohort D.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2023-10-07 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) determined by the researchers according to the RECIST 1.1 criteria.. | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Progression-free survival (PFS) is defined as the time from the date of the first dose to the earlier of the dates of the first objective documentation of radiographic progressive disease (PD) or death due to any cause.

SECONDARY OUTCOMES:
Overall survival | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Overall survival (OS) is defined as the time from the date of first dose to the date of death from any cause.
Overall response rate | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Objective response rate (defined as CR+PR) will be reported based on investigator's evaluation.
Disease control rate | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Disease control rate (defined as CR+PR+SD) will be reported based on investigator's evaluation.
Duration of response | Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever occurs first), up to 24 months post-dose
  Duration of response (DOR) is defined as the time from the date of the first response to the first objective documentation of radiographic progressive disease (PD) or death due to any cause.
Treatment-related adverse event | Informed consent to 30 days after last dose of treatment
  A treatment-related adverse event (TRAE) is defined as any adverse event not present prior to the initiation of drug treatment or any adverse event already present that worsens in intensity or frequency following exposure to the drug treatment. TRAEs were graded using National Cancer Institute (NCI)-CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: zhenghang Wang, Study Director — Peking University Cancer Hospital & Institute
Locations (10):
- China (10):
  - Department of Gastrointestinal Oncology, Key Laboratory of Carcinogenesis and Translational Research (Ministry of Education), Peking University Cancer Hospital & Institute, Beijin, Beijing Municipality
  - Department of Gastroenterology and Hepatology, The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Department of Oncology, The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Medical Oncology Department of Gastrointestinal Cancer, Liaoning Cancer Hospital & Institute, Shengyang, Liaoning
  - Department of Oncology, The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Department of Gastroenterology, Shanxi Province Cancer Hospital/Shanxi Hospital Affiliated to Cancer Hospital, Taiyuan, Shanxi
  - Department of Medical Oncology, Peking University First Hospital, Beijing
  - Department of Oncology, Beijing Luhe Hospital Affiliated to Capital Medical University, Beijing
  - Department of Oncology, Peking University Shougang Hospital, Beijing
  - Department of Gastrointestinal Oncology, Tianjin Medical University Cancer Institute and Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luchini C, Bibeau F, Ligtenberg MJL, Singh N, Nottegar A, Bosse T, Miller R, Riaz N, Douillard JY, Andre F, Scarpa A. ESMO recommendations on microsatellite instability testing for immunotherapy in cancer, and its relationship with PD-1/PD-L1 expression and tumour mutational burden: a systematic review-based approach. Ann Oncol. 2019 Aug 1;30(8):1232-1243. doi: 10.1093/annonc/mdz116. PMID 31056702
- [Background] Le DT, Durham JN, Smith KN, Wang H, Bartlett BR, Aulakh LK, Lu S, Kemberling H, Wilt C, Luber BS, Wong F, Azad NS, Rucki AA, Laheru D, Donehower R, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Greten TF, Duffy AG, Ciombor KK, Eyring AD, Lam BH, Joe A, Kang SP, Holdhoff M, Danilova L, Cope L, Meyer C, Zhou S, Goldberg RM, Armstrong DK, Bever KM, Fader AN, Taube J, Housseau F, Spetzler D, Xiao N, Pardoll DM, Papadopoulos N, Kinzler KW, Eshleman JR, Vogelstein B, Anders RA, Diaz LA Jr. Mismatch repair deficiency predicts response of solid tumors to PD-1 blockade. Science. 2017 Jul 28;357(6349):409-413. doi: 10.1126/science.aan6733. Epub 2017 Jun 8. PMID 28596308
- [Background] Wang Z, Zhao X, Gao C, Gong J, Wang X, Gao J, Li Z, Wang J, Yang B, Wang L, Zhang B, Zhou Y, Wang D, Li X, Bai Y, Li J, Shen L. Plasma-based microsatellite instability detection strategy to guide immune checkpoint blockade treatment. J Immunother Cancer. 2020 Nov;8(2):e001297. doi: 10.1136/jitc-2020-001297. PMID 33172882
- [Background] Andre T, Shiu KK, Kim TW, Jensen BV, Jensen LH, Punt C, Smith D, Garcia-Carbonero R, Benavides M, Gibbs P, de la Fouchardiere C, Rivera F, Elez E, Bendell J, Le DT, Yoshino T, Van Cutsem E, Yang P, Farooqui MZH, Marinello P, Diaz LA Jr; KEYNOTE-177 Investigators. Pembrolizumab in Microsatellite-Instability-High Advanced Colorectal Cancer. N Engl J Med. 2020 Dec 3;383(23):2207-2218. doi: 10.1056/NEJMoa2017699. PMID 33264544
- [Background] Zhu M, Jin Z, Hubbard JM. Management of Non-Colorectal Digestive Cancers with Microsatellite Instability. Cancers (Basel). 2021 Feb 6;13(4):651. doi: 10.3390/cancers13040651. PMID 33561950
- [Background] Chida K, Kawazoe A, Kawazu M, Suzuki T, Nakamura Y, Nakatsura T, Kuwata T, Ueno T, Kuboki Y, Kotani D, Kojima T, Taniguchi H, Mano H, Ikeda M, Shitara K, Endo I, Yoshino T. A Low Tumor Mutational Burden and PTEN Mutations Are Predictors of a Negative Response to PD-1 Blockade in MSI-H/dMMR Gastrointestinal Tumors. Clin Cancer Res. 2021 Jul 1;27(13):3714-3724. doi: 10.1158/1078-0432.CCR-21-0401. Epub 2021 Apr 29. PMID 33926917
- [Background] Wang Z, Wang X, Xu Y, Li J, Zhang X, Peng Z, Hu Y, Zhao X, Dong K, Zhang B, Gao C, Zhao X, Chen H, Cai J, Bai Y, Sun Y, Shen L. Mutations of PI3K-AKT-mTOR pathway as predictors for immune cell infiltration and immunotherapy efficacy in dMMR/MSI-H gastric adenocarcinoma. BMC Med. 2022 Apr 21;20(1):133. doi: 10.1186/s12916-022-02327-y. PMID 35443723
- [Background] Wang Z, Zhang Q, Qi C, Bai Y, Zhao F, Chen H, Li Z, Wang X, Chen M, Gong J, Peng Z, Zhang X, Cai J, Chen S, Zhao X, Shen L, Li J. Combination of AKT1 and CDH1 mutations predicts primary resistance to immunotherapy in dMMR/MSI-H gastrointestinal cancer. J Immunother Cancer. 2022 Jun;10(6):e004703. doi: 10.1136/jitc-2022-004703. PMID 35705314
- [Background] Malla M, Loree JM, Kasi PM, Parikh AR. Using Circulating Tumor DNA in Colorectal Cancer: Current and Evolving Practices. J Clin Oncol. 2022 Aug 20;40(24):2846-2857. doi: 10.1200/JCO.21.02615. Epub 2022 Jul 15. PMID 35839443
- [Background] Zhang Q, Luo J, Wu S, Si H, Gao C, Xu W, Abdullah SE, Higgs BW, Dennis PA, van der Heijden MS, Segal NH, Chaft JE, Hembrough T, Barrett JC, Hellmann MD. Prognostic and Predictive Impact of Circulating Tumor DNA in Patients with Advanced Cancers Treated with Immune Checkpoint Blockade. Cancer Discov. 2020 Dec;10(12):1842-1853. doi: 10.1158/2159-8290.CD-20-0047. Epub 2020 Aug 14. PMID 32816849
- [Background] Kasi PM, Budde G, Krainock M, Aushev VN, Koyen Malashevich A, Malhotra M, Olshan P, Billings PR, Aleshin A. Circulating tumor DNA (ctDNA) serial analysis during progression on PD-1 blockade and later CTLA-4 rescue in patients with mismatch repair deficient metastatic colorectal cancer. J Immunother Cancer. 2022 Jan;10(1):e003312. doi: 10.1136/jitc-2021-003312. PMID 35101943
- [Background] Luo J, Wu S, Rizvi H, Zhang Q, Egger JV, Osorio JC, Schoenfeld AJ, Plodkowski AJ, Ginsberg MS, Callahan MK, Maher C, Shoushtari AN, Postow MA, Voss MH, Kotecha RR, Gupta A, Raja R, Kris MG, Hellmann MD. Deciphering radiological stable disease to immune checkpoint inhibitors. Ann Oncol. 2022 Aug;33(8):824-835. doi: 10.1016/j.annonc.2022.04.450. Epub 2022 May 6. PMID 35533926
- [Background] Bui QL, Mas L, Hollebecque A, Tougeron D, de la Fouchardiere C, Pudlarz T, Alouani E, Guimbaud R, Taieb J, Andre T, Colle R, Cohen R. Treatments after Immune Checkpoint Inhibitors in Patients with dMMR/MSI Metastatic Colorectal Cancer. Cancers (Basel). 2022 Jan 14;14(2):406. doi: 10.3390/cancers14020406. PMID 35053568
- [Background] Hollebecque A, Chung HC, de Miguel MJ, Italiano A, Machiels JP, Lin CC, Dhani NC, Peeters M, Moreno V, Su WC, Chow KH, Galvao VR, Carlsen M, Yu D, Szpurka AM, Zhao Y, Schmidt SL, Gandhi L, Xu X, Bang YJ. Safety and Antitumor Activity of alpha-PD-L1 Antibody as Monotherapy or in Combination with alpha-TIM-3 Antibody in Patients with Microsatellite Instability-High/Mismatch Repair-Deficient Tumors. Clin Cancer Res. 2021 Dec 1;27(23):6393-6404. doi: 10.1158/1078-0432.CCR-21-0261. Epub 2021 Aug 31. PMID 34465599
- [Background] Chen M, Wang Z, Liu Z, Liu N, Fang W, Zhang H, Jin X, Li J, Zhao W, Qu H, Song F, Chang Z, Li Y, Tang Y, Xu C, Zhang X, Wang X, Peng Z, Cai J, Li J, Shen L. The Optimal Therapy after Progression on Immune Checkpoint Inhibitors in MSI Metastatic Gastrointestinal Cancer Patients: A Multicenter Retrospective Cohort Study. Cancers (Basel). 2022 Oct 21;14(20):5158. doi: 10.3390/cancers14205158. PMID 36291942